CLINICAL TRIAL: NCT02048124
Title: Prospective Study Comparing the Diagnostic Yield of Solid Lesion Biopsies Performed by EUS-FNA Using the 25d ProCor Needle Versus the Standard 25g Needle.
Brief Title: Study Comparing 25d ProCor Needle Versus the Standard 25g Needle for Biopsies Performed by EUS-FNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CE 13.030
Record Dates: First submitted 2014-01-09; First posted 2014-01-29 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-05

CONDITIONS: Solid Lesion Biopsies
Keywords: 25d ProCor needle; 22 gauge; endoscopic ultrasonography; fine needle biopsies; Patients; presenting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 25g standard needle (Active Comparator): EUS-FNA passes will be performed without stylet. One "needle pass" is defined as 5 strokes in 4 different areas of the lesion. The material from the needle passes will be expressed into formalin to look for core samples. Material from the next needle passes will be expressed onto slides for cytological analysis. Ease of puncture will be scored qualitatively as poor (scored 1), good (scored 2) or excellent (scored 3).
  Interventions: Device: 25g standard needle
- 25d ProCor needle (Experimental): EUS-FNA passes will be performed without stylet. One "needle pass" is defined as 5 strokes in 4 different areas of the lesion. The material from the needle passes will be expressed into formalin to look for core samples. Material from the next needle passes will be expressed onto slides for cytological analysis. Ease of puncture will be scored qualitatively as poor (scored 1), good (scored 2) or excellent (scored 3).
  Interventions: Device: 25d ProCor needle

INTERVENTIONS:
Device: 25g standard needle
  Other Names: Evaluation of core samples; Cytological analysis; Ease of puncture
  Arms: 25g standard needle
Device: 25d ProCor needle
  Arms: 25d ProCor needle

SUMMARY:
Background: There is an ongoing interest in developing Endoscopic Ultrasound /Fine Needle Aspiration (EUS-FNA) needles that can provide tissue core biopsies for a true histological (rather than cytological) evaluation. By slightly modifying the traditional EUS-FNA needle, a new needle named "ProCor" was developed in the hope of obtaining core samples and thus increase diagnostic yield.

Objective: In this research project, we propose to conduct a prospective trial to compare the results obtained with two types of needles: a 25g standard needle (25gS) and the 25g ProCor needle (25gP).

EUS-FNA Biopsies will be obtained with both the 25S and 25P needles in each lesion; a randomisation sequence will set in order to determine which of the two needles will first be used (25S or 25P).

The cytological or histological diagnoses will be made; . for histological diagnosis, the pathologist will first establish the presence or absence of a tissue core (defined as a measurable cylinder of tissue). The pathologist will assess the adequacy of each specimen: cellularity (score 1 "poor"; score 2 "good"; score 3 "excellent"),[14] sample bloodiness (score 1 "minimal";score 2 "moderate"; score 3 "significant", and the presence or absence of malignancy("positive" / "negative" / "suspicious" / inconclusive).

Results for continuous variables will be summarized using mean ± SD, . and categorical variables using proportions. The 25S and 25P groups will be compared using Chi-square test for categorical variables and, Student t test for continuous variablesTwo-sided p values less than 0.05 will be considered statistically significant. Data will be analyzed using SPSS v 15.0 (SPSS Inc., Chicago IL) statistical software.

DETAILED DESCRIPTION:
Objectives of the study

The primary objective is to compare the diagnostic yield of biopsies performed by EUS-FNA using the 25d ProCor needle versus the standard 25g needle.

The primary outcome is the diagnostic yield defined as: sensitivity for the presence of cancer based on the analysis of EUS-FNA samples.

The secondary objectives are:

1. to compare the size of the "core" samples produced by the two types of needles.
2. to compare the incidence and severity of immediate complications associated with the two types of needles

Methods

Design: This a prospective clinical study for the validation of a new instrument (ProCor biopsy needle) for application to clinical medicine, namely the diagnosis of cancer.

Endoscopic procedures:

Informed consent by the patient will be obtained before each procedure by a single research assistant.

All EUS examinations will be performed under conscious sedation (midazolam, fentanyl) by one two experienced endosonographers according to the standard procedures at the CHUM and using a linear echoendoscope. , If the lesion is considered solid and EUS-FNA is considered clinically indicated and safe, the patient will be enrolled and the randomisation envelope will be opened. EUS-FNA Biopsies will be obtained with both the 25S and 25P needles in each lesion; a randomisation sequence will set in order to determine which of the two needles will first be used (25S or 25P).

EUS-FNA passes will be performed without stylet. One "needle pass" is defined as 5 strokes in 4 different areas of the lesion. The material from the first 2 needle passes (one 25S and the other 25P) will be expressed into formalin to look for core samples. Material from the next 2 needle passes (again one 25S and the other 25P) will be expressed onto slides for cytological analysis. Ease of puncture will be scored qualitatively as poor (scored 1), good (scored 2) or excellent (scored 3).

Immediate complications will be assessed and recorded by nurses and/or physicians during the procedure as well after the procedure while the patients will be monitored in the recovery room for at least 60 minutes before discharge.

The areas which will be investigated by biopsy will be the pancreas, the retroperitoneal and/or the mediastinal lymph nodes.

Cytological and Histological analyses:

Samples from all needle passes will be stained using a standard Papanicolaou stain and analyzed by one experienced pathologist who will be blinded as to needle type. The cytological or histological diagnoses will be made; . for histological diagnosis, the pathologist will first establish the presence or absence of a tissue core (defined as a measurable cylinder of tissue). The pathologist will assess the adequacy of each specimen: cellularity (score 1 "poor"; score 2 "good"; score 3 "excellent"),[14] sample bloodiness (score 1 "minimal";score 2 "moderate"; score 3 "significant", and the presence or absence of malignancy("positive" / "negative" / "suspicious" / inconclusive).

Diagnostic yield Diagnostic yield is defined as sensitivity for the presence of cancer based on the analysis of EUS-FNA samples. The gold standard will be the presence of cancer as defined on the basis of at least one of the following two criteria: positive cytological or histological results and malignant disease after clinical follow up (clinical worsening and radiologic evidence of progression within the 6 months following FNA).

Data collection

Clinical data will be collected prospectively and saved in a database. In addition to demographics, these will include:

* size and location (pancreas, lymph node, liver, adrenal gland, others) of the target lesion
* technical and procedure variables ( FNA path, , number of needle passes, needle visibility, ease to puncture, needle failure, cellularity, bloodiness)
* cytological diagnosis
* final diagnosis
* immediate complications. Research data and project-related documents will be preserved during 15 year after the end of the study.

Statistical analysis Results for continuous variables will be summarized using mean ± (Standard Deviation) SD, . and categorical variables using proportions. The 25S and 25P groups will be compared using Chi-square test for categorical variables and, Student t test for continuous variablesTwo-sided p values less than 0.05 will be considered statistically significant. Data will be analyzed using SPSS v 15.0 (SPSS Inc., Chicago IL) statistical software.

Sample size The sample size is calculated as a study of non-inferiority. Assuming a sensitivity for cancer of 85% for the 25S needle and a difference of sensitivity of 15% as clinically significant, a sample size of 112 patients per group would be needed (α = 0.05 and β = 0.2). Since we perform approximately 400 EUS-FNA biopsies for solid lesions annually,. it is expected that this study could be completed within approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old
* Patients presenting with a solid lesion
* Patients for whom EUS-FNA is considered clinically indicated and safe

Exclusion Criteria:

* Age < 18 years old,
* Patients with suspected diagnosis of lymphoma, GIST, sarcoidosis or other lesions in which a large amount of tissue will be required for diagnosis,
* Patients with significant coagulopathy (INR>1.5, platelets <50000/mm3, use of low molecular weight heparin, use of clopidogrel within 7 days of EUS), Patients presenting with cystic lesions Inability or refusal to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Compare the diagnostic yield of biopsies performed EUS-FNA by using the 25d ProCor needle versus the standard 25g needle | 1 day

SECONDARY OUTCOMES:
Measurement of the size of the "core" samples produced by the two types of needles | 1 day
Measurement of incidence and severity of immediate complications associated with the two types of needles | 1 day
  Immediate complications will be assessed and recorded by nurses and/or physicians during and after the procedure while the patient was recovering from sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Anand V Sahai, MD, Principal Investigator — Hopital Saint Luc (Centre Hopitalier de l´Université du Montreal) Montreal, Quebec, Canada
Locations (1):
- Hopital Saint Luc (Centre Hopitalier de l´Université du Montreal), Montreal, Quebec, Canada

REFERENCES:
- [Background] Crowe DR, Eloubeidi MA, Chhieng DC, Jhala NC, Jhala D, Eltoum IA. Fine-needle aspiration biopsy of hepatic lesions: computerized tomographic-guided versus endoscopic ultrasound-guided FNA. Cancer. 2006 Jun 25;108(3):180-5. doi: 10.1002/cncr.21912. PMID 16634071
- [Background] Nguyen P, Feng JC, Chang KJ. Endoscopic ultrasound (EUS) and EUS-guided fine-needle aspiration (FNA) of liver lesions. Gastrointest Endosc. 1999 Sep;50(3):357-61. doi: 10.1053/ge.1999.v50.97208. PMID 10462656
- [Background] Jenssen C, Dietrich CF. Endoscopic ultrasound-guided fine-needle aspiration biopsy and trucut biopsy in gastroenterology - An overview. Best Pract Res Clin Gastroenterol. 2009;23(5):743-59. doi: 10.1016/j.bpg.2009.05.006. PMID 19744637
- [Background] Paquin SC, Gariepy G, Lepanto L, Bourdages R, Raymond G, Sahai AV. A first report of tumor seeding because of EUS-guided FNA of a pancreatic adenocarcinoma. Gastrointest Endosc. 2005 Apr;61(4):610-1. doi: 10.1016/s0016-5107(05)00082-9. No abstract available. PMID 15812422
- [Background] Eloubeidi MA, Chen VK, Eltoum IA, Jhala D, Chhieng DC, Jhala N, Vickers SM, Wilcox CM. Endoscopic ultrasound-guided fine needle aspiration biopsy of patients with suspected pancreatic cancer: diagnostic accuracy and acute and 30-day complications. Am J Gastroenterol. 2003 Dec;98(12):2663-8. doi: 10.1111/j.1572-0241.2003.08666.x. PMID 14687813
- [Background] Savides TJ, Donohue M, Hunt G, Al-Haddad M, Aslanian H, Ben-Menachem T, Chen VK, Coyle W, Deutsch J, DeWitt J, Dhawan M, Eckardt A, Eloubeidi M, Esker A, Gordon SR, Gress F, Ikenberry S, Joyce AM, Klapman J, Lo S, Maluf-Filho F, Nickl N, Singh V, Wills J, Behling C. EUS-guided FNA diagnostic yield of malignancy in solid pancreatic masses: a benchmark for quality performance measurement. Gastrointest Endosc. 2007 Aug;66(2):277-82. doi: 10.1016/j.gie.2007.01.017. PMID 17643700
- [Background] Williams DB, Sahai AV, Aabakken L, Penman ID, van Velse A, Webb J, Wilson M, Hoffman BJ, Hawes RH. Endoscopic ultrasound guided fine needle aspiration biopsy: a large single centre experience. Gut. 1999 May;44(5):720-6. doi: 10.1136/gut.44.5.720. PMID 10205212
- [Background] Wang KX, Ben QW, Jin ZD, Du YQ, Zou DW, Liao Z, Li ZS. Assessment of morbidity and mortality associated with EUS-guided FNA: a systematic review. Gastrointest Endosc. 2011 Feb;73(2):283-90. doi: 10.1016/j.gie.2010.10.045. PMID 21295642